CLINICAL TRIAL: NCT02572674
Title: Study of Predictor of Mood Relapse in Bipolar Disorders : Prospective, Clinical, Neuropsychological, Biological and Genetic Study
Brief Title: Study of Predictor of Mood Relapse in Bipolar Disorders
Acronym: RechuteBP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P071245
Record Dates: First submitted 2015-08-13; First posted 2015-10-09 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Bipolar Disorder; Euthymic State
Keywords: Bipolar disorder; relapse risk factors; prospective follow up
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- experimental arm (Other): Experimental follow up : Neuropsychological assessment at 6 month and genetic samples
  Interventions: Other: Experimental follow up; Genetic: Genetic sample

INTERVENTIONS:
Other: Experimental follow up — Neuropsychological assessment (intellectual functioning, episodic verbal memory, processing speed, attention, working verbal memory, working visual memory, executive function)
Genetic: Genetic sample — Blood samples

SUMMARY:
Study in 400 patients with bipolar disorder I or II, of relapse risk factors. The principal objective of this research is to test the predictive value of core vulnerability dimensions such as affective instability and emotional reactivity, measured by validated questionnaires (AIM and ALS) on recurrence of affective major episode (depressed, hypomanic or manic) during a 24 months prospective follow-up.

In addition, several arguments suggest that inter-individual variability in the risk of relapse is influenced by genetic factors. In particular, the implication of such factors have been demonstrated in rapid cycling or antidepressants induced mania. However, this has never been tested in cohorts followed prospectively. Finally, the existence of neuropsychological deficits in bipolar disorder is well documented and their role in the risk of relapse is suspected. Yet the nature of these deficits, their origin and evolutionary course remain poorly investigated. In summary, the secondary objectives of this research are the study of the influence of these other clinical, neuropsychological and genetic factors on the risk of relapse.

• Scientific rationale The dimensions of affective instability and emotional reactivity, are considered core psychological and temperamental vulnerability dimensions to bipolar disorder. Differences in levels of instability and reactivity may account for the inter-individual variability observed in bipolar disorder in terms of risk of relapse. These dimensions are measured using validated questionnaires (Affective Instability Measure (AIM) and Affective Lability Scale (ALS)). Relapsing is defined as the occurrence of a depressive episode, hypomanic, manic or mixed episode (DSMIV criteria).

Other factors that may influence the risk of relapse have been suggested in the literature but have not been formally tested in prospective studies:

1. cognitive deficits: the existence of neuropsychological deficits in bipolar disorder are well documented and their role in the risk of relapse is suspected. Yet the nature of these deficits, their origin and their course remain poorly investigated. Indeed, some appear to be related to the neurotoxicity of the episodes themselves, the other being related to the vulnerability to bipolar disorder
2. The involvement of genetic vulnerability factors in bipolar disorder is widely demonstrated. Several arguments suggest the implication of genetic factors in the risk of relapse. This is the case for some outcome patterns such as rapid cycling or antidepressants induced mania. Again, this has never been tested in cohorts followed prospectively.
3. The role of certain inflammatory and infectious factors in the etiology of bipolar disorder has been suggested but it is clear whether these biomarkers are "state" or "traits". Thus, the role of neurotoxic inflammatory or infectious factors in relapse mood has never been tested in a prospective follow up studies.

   * Main objective of the project To determine if the scores of AIM and ALS, assessed at baseline in euthymic bipolar patients is associated with relapse in patients during a 2 years follow-up period.
   * Secondary objectives of the project Determine if the neuropsychological performance at T0, measured in euthymic patients predict relapse during a 2 years follow-up period.

Determine whether the neuropsychological deficits observed in euthymic bipolar patients that contribute to functional impairment worsen with time.

DNA collection to test the involvement of candidate genes Serum collection to study the biological and infectious biomarkers

• Methodology Prospective follow up studies. Multicenter.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar disorder I or II
* French language
* Aging between 18 years and 55 years
* Young Mania Rating Scale (YMRS) < 12
* Montgomery Asberg Depression Rating Scale (MDRS) < 10

Exclusion Criteria:

* Rapid cycling
* Undefined number of major relapses
* Drug and alcohol abuse within 6 months
* Electroconvulsive therapy (ECT) within 12 months
* Epilepsy, traumatism cranial or other neurological diseases
* Daltonism or visual trouble

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 274 (Actual)
Dates: Start 2010-05; Primary Completion 2016-08 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Combined outcome based on AIM and ALS's score assessed at baseline in euthymic bipolar patients associated with relapse in patients during a 2 years follow-up period. | 24 months

SECONDARY OUTCOMES:
Global neuropsychological performance based on combined score of all neuropsychological scales (detail below) at T0, measured in euthymic patients predict relapse during a 2 years follow-up period. | 24 months
  Neuropsychological scales : intellectual functioning, episodic verbal memory, processing speed, attention, working verbal memory, working visual memory, executive function
Global neuropsychological deficits based on combined score of all neuropsychological scales (detail below) observed in euthymic bipolar patients that contribute to functional impairment worsen with time | 24 months
  Neuropsychological scales : intellectual functioning, episodic verbal memory, processing speed, attention, working verbal memory, working visual memory, executive function

CONTACTS AND LOCATIONS:
Overall Officials: Frank BELLIVIVIER, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Fernand Widal Hospital, Paris, France